CLINICAL TRIAL: NCT00737464
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous MIRCERA for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Once Monthly Intravenous Mircera for the Maintenance Treatment of Dialysis Patients With Chronic Renal Anemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21810
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mircera (Experimental): Participant with chronic renal anemia will receive methoxy polyethylene glycol-epoetin beta [Mircera] intravenously (IV) [(120, 200 or 360 micrograms (mcg)] every 4 weeks for 12 weeks.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — iv (120, 200 or 360 micrograms) every 4 weeks for 12 weeks.

SUMMARY:
This single arm study will evaluate the maintenance of hemoglobin levels, safety and tolerability of once-monthly intravenous administration of Mircera in dialysis patients with chronic renal anemia. Patients will receive intravenous Mircera (120, 200 or 360 micrograms) every four weeks depending on the previous dose of epoetin alfa administered in the week preceding first study drug administration. Patients will be treated for 12 weeks with follow up 2 weeks after the last treatment visit. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, >=18 years of age;
* chronic renal anemia;
* Hb concentration 10.5g/dL - 12.5g/dL;
* continuous intravenous maintenance therapy with epoetin alfa at the same dosing interval during the previous 2 months.

Exclusion Criteria:

* blood transfusion within the previous 2 months;
* poorly controlled hypertension;
* significant acute or chronic bleeding;
* active malignant disease;
* congestive heart failure (NYHA Class IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-08-26 (Actual); Primary Completion 2009-09-12 (Actual); Study Completion 2009-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- India (17):
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Manipal Institute of Nephrology and Urology; Nephrology, Bangalore
  - Columbia Asia Medical Centre - Hebbal; Nephrology, Bangalore
  - Tanker Foundation, Chennai
  - MIOT Institute of Nephrology ; Nephrology, Chennai
  - Madras Medical Mission Hospital, Chennai
  - International Hospital, Guwahati
  - Kamineni Hospitals; Nephrology, Hyderabad
  - Nizam's Institute of Medical Sciences; Nephrology, Hyderabad
  - Regency Hospital Ltd.; Nephrology, Kanpur
  - Wockhardt Hospital and Kidney Institute; Nephrology, Kolkata
  - Meerut Kidney Hospital, Meerut
  - Silver Oaks Hospital; Nephrology, Mohali
  - Apex Kidney Care, Mumbai
  - Lancelot Dialysis Center, Mumbai
  - Fortis Flt. Lt. Rajan Dhall Hospital; Nephrology, New Delhi
  - Ruby Hall Clinic, Pune

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 participants were enrolled from 26 August 2008 to 12 September 2009 at 11 study sites in India.
Groups:
- Mircera: Eligible participants with chronic renal anemia were administered methoxy polyethylene glycol-epoetin beta [Mircera] intravenously (IV) [(120, 200 or 360 micrograms (mcg)] every 4 weeks for 12 weeks.
Period: Overall Study
Arm/Group | Mircera
Started | 132
Completed | 114
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Death | 6
Not completed — Other - Failure to Return | 1
Not completed — Refused Treatment / Withdrew Consent | 6
Not completed — Other reasons | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of study medication.
Arm/Group | Mircera
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.74 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 97

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Mean Hemoglobin Levels Within the Target Range During the Last 4 Weeks of the Treatment Period (Weeks 8 to 12)
Description: Participants maintaining mean hemoglobin (Hb) concentration within the target range i.e. 10.0 - 12.0 gram per deciliter (g/dL) during last 4 weeks (Weeks 8 to 12) of treatment period (TP) were reported. Total duration for treatment period was 12 weeks. Stability verification period of 2-weeks was conducted before treatment period. The reference Hb concentrations were based upon the mean of the assessments at Weeks -2, -1 and Week 0. The target range for assessment was set at the reference value Hb +/- 1 g/dL but not >12.0 g/dL and not <10.0 g/dL.
Time Frame: Weeks 8 to 12 (Last 4 weeks of treatment period)
Population: Per-protocol (PP) population comprised of participants who had received at least 1 dose of MIRCERA (Week 0) and for whom data for at least one follow-up variable was available and who had completed the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Mircera: Eligible participants were administered methoxy polyethylene glycol-epoetin beta [Mircera] intravenously (IV) [(120, 200 or 360 micrograms (mcg)] every 4 weeks for 12 weeks.
Arm/Group | Mircera
Number analyzed (Participants) | 114
Percentage of participants | 57.89 [48.29 to 67.08]

2. Secondary Outcome: Mean Hemoglobin Concentration Between Stability Verification Period (Weeks -2 to -1) and Treatment Period (Weeks 8 to 12)
Description: The mean change in Hb concentration between reference stability verification period (SVP) and in last 4 weeks (Weeks 8 to 12) of treatment period (TP) was reported. Duration for SVP was 2 weeks followed by treatment period of 12 weeks. The reference Hb concentrations were based upon the mean of the assessments at Weeks -2, -1 and Week 0. The target range for assessment was set at the reference value hemoglobin +/- 1 g/dL but not >12.0 g/dL and not <10.0 g/dL.
Time Frame: SVP (Weeks -2 to -1) and TP (Weeks 8 to 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Mircera
Number analyzed (Participants) | 114
gm/dL
  Hb in SVP | 10.76 (0.75)
  Avg of Hb in Last 4 Weeks TP | 11.28 (1.22)
Statistical Analysis 1: Comparison: Mircera; Test type: Superiority or Other; Mean Difference (Final Values) = 0.52

3. Secondary Outcome: Mean Time Participants Spent Having Hemoglobin Range of 10.0 to 12.0 g/dL
Description: Mean time participants spent having hemoglobin range of 10.0 to 12.0 g/dL was reported. The reference Hb concentrations were based upon the mean of the assessments at Weeks -2, -1 and Week 0. The target range for assessment was set at the reference value hemoglobin +/- 1 gram per deciliter but not >12.0 g/dL and not <10.0 g/dL.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Mircera
Number analyzed (Participants) | 114
Weeks | 3.15 (1.00)

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events, Serious Adverse Events and Deaths
Description: Participants with treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and deaths in the overall study were reported. An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 14
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | Mircera
Number analyzed (Participants) | 132
Number of participants
  TEAEs | 27
  SAEs | 9
  Deaths | 3

5. Secondary Outcome: Mean Change From Baseline in Heart Rate Over Time
Description: Mean change from Baseline (Week -1) to end of the treatment (Week 12) in heart rate was reported. Baseline measure was considered as (Week -1) evaluation for this parameter.
Time Frame: From Baseline (Week -1) to Weeks 0, 1, 2, 4, 6, 8, 10, and 12
Population: Safety population included all enrolled participants who received at least one dose of study drug. n = number of participants analyzed at a given time point.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Mircera
Number analyzed (Participants) | 132
Beats per minute (bpm)
  Heart rate, Week -1, (n = 132) | 78.79 (7.12)
  Heart rate, Week 0, (n = 131) | 79.54 (7.27)
  Heart rate, Week 1, (n = 129) | 78.64 (6.92)
  Heart rate, Week 2, (n = 124) | 78.98 (7.83)
  Heart rate, Week 4, (n = 124) | 78.61 (6.92)
  Heart rate, Week 6, (n = 121) | 79.55 (8.37)
  Heart rate, Week 8, (n = 118) | 79.83 (7.55)
  Heart rate, Week 10, (n = 115) | 79.56 (7.54)
  Heart rate, Week 12, (n = 115) | 79.80 (7.65)

6. Secondary Outcome: Mean Change From Baseline in Blood Pressure (Systolic Blood Pressure and Diastolic Blood Pressure) Over Time
Description: Mean change from Baseline (Week -2) to end of the treatment (Week 12) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) before and after dialysis was reported. Baseline measure was considered as (Week -2) evaluation for this parameter.
Time Frame: From Baseline (Week -2) to Weeks -1, 0, 1, 2, 4, 6, 8, 10, and 12
Population: Safety population included all enrolled participants who received at least one dose of study drug. n = the number of participants analyzed at a given time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mircera
Number analyzed (Participants) | 132
mmHg
  SBP, Week-2, Before Dialysis (n = 132) | 145.04 (15.71)
  SBP, Week-2, After Dialysis (n = 131) | 145.51 (18.12)
  SBP, Week-1, Before Dialysis (n = 132) | 146.72 (14.77)
  SBP, Week-1, After Dialysis (n =131) | 143.26 (18.72)
  SBP, Week 0, Before Dialysis (n = 131) | 145.05 (16.04)
  SBP, Week 0, After Dialysis (n = 130) | 143.75 (16.96)
  SBP, Week 1, Before Dialysis (n = 129) | 147.02 (17.40)
  SBP, Week 1, After Dialysis (n = 128) | 144.02 (17.68)
  SBP, Week 2, Before Dialysis (n = 124) | 146.85 (18.08)
  SBP, Week 2, After Dialysis (n = 123) | 144.92 (18.44)
  SBP, Week 4, Before Dialysis (n = 124) | 146.68 (16.98)
  SBP, Week 4, After Dialysis (n = 124) | 143.65 (18.18)
  SBP, Week 6, Before Dialysis (n = 121) | 145.16 (18.58)
  SBP, Week 6, After Dialysis (n = 121) | 145.55 (20.64)
  SBP, Week 8, Before Dialysis (n = 118) | 144.77 (18.84)
  SBP, Week 8, After Dialysis (n = 118) | 143.42 (17.14)
  SBP, Week 10, Before Dialysis (n = 115) | 144.14 (17.57)
  SBP, Week 10, After Dialysis (n = 115) | 143.98 (17.44)
  SBP, Week 12, Before Dialysis (n = 115) | 144.55 (18.46)
  SBP, Week 12, After Dialysis (n = 115) | 143.80 (18.22)
  DBP, Week -2, Before Dialysis (n = 132) | 82.92 (9.32)
  DBP, Week -2, After Dialysis (n = 131) | 84.05 (9.40)
  DBP, Week -1, Before Dialysis (n = 132) | 83.90 (9.80)
  DBP, Week -1, After Dialysis (n = 131) | 83.22 (9.51)
  DBP, Week 0, Before Dialysis (n = 131) | 84.05 (8.57)
  DBP, Week 0, After Dialysis (n = 130) | 84.04 (8.94)
  DBP, Week 1, Before Dialysis (n = 129) | 84.68 (9.34)
  DBP, Week 1, After Dialysis (n = 128) | 83.27 (8.97)
  DBP, Week 2, Before Dialysis (n = 124) | 83.77 (8.62)
  DBP, Week 2, After Dialysis (n = 123) | 83.69 (8.85)
  DBP, Week 4, Before Dialysis (n = 124) | 84.15 (8.98)
  DBP, Week 4, After Dialysis (n = 124) | 83.29 (9.27)
  DBP, Week 6, Before Dialysis (n = 121) | 83.31 (8.98)
  DBP, Week 6, After Dialysis (n = 121) | 83.97 (9.24)
  DBP, Week 8, Before Dialysis (n = 118) | 83.28 (9.49)
  DBP, Week 8, After Dialysis (n = 118) | 84.35 (8.03)
  DBP, Week 10, Before Dialysis (n = 115) | 83.91 (8.55)
  DBP, Week 10, After Dialysis (n = 115) | 84.33 (9.24)
  DBP, Week 12, Before Dialysis (n = 115) | 84.17 (10.47)
  DBP, Week 12, After Dialysis (n = 115) | 83.23 (9.45)

7. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram
Description: Participants with abnormal electrocardiogram were reported.
Time Frame: At Week -2 and Week 12
Population: as for outcome 6
Measure: Number; unit: Number of participants
Arm/Group | Mircera
Number analyzed (Participants) | 132
Number of participants
  Week -2 (n=132) | 61
  Week 12 (n=115) | 50

8. Secondary Outcome: Mean Values of White Blood Cells and Platelets Over Time
Description: Mean values of white blood cells (WBCs), and platelets at Weeks -2, 4, 8, and 12 were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Per cubic millimeter
Arm/Group | Mircera
Number analyzed (Participants) | 132
Per cubic millimeter
  WBCs, Week -2 (n = 132) | 7527.50 (2444.43)
  WBCs, Week 4 (n = 114) | 7369.74 (2470.21)
  WBCs, Week 8 (n = 118) | 7506.61 (2214.38)
  WBCs, Week 12 (n = 115) | 7484.35 (2130.22)
  Platelets, Week -2 (n = 132) | 211772.73 (73360.93)
  Platelets, Week 4 (n = 114) | 199508.77 (64724.91)
  Platelets, Week 8 (n = 118) | 208745.76 (67546.15)
  Platelets, Week 12 (n = 115) | 208566.37 (102269.07)

9. Secondary Outcome: Mean Values of Hypochromic Red Blood Cells Over Time
Description: Mean values of hypochromic red blood cells (RBCs) at Weeks -2, 4, 8, and 12 were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of RBCs
Arm/Group | Mircera
Number analyzed (Participants) | 42
Percentage of RBCs
  Hypochromic RBCs, Week -2 (n = 41) | 3.58 (0.43)
  Hypochromic RBCs, Week 4 (n = 34) | 3.73 (0.57)
  Hypochromic RBCs, Week 8 (n = 42) | 3.88 (0.59)
  Hypochromic RBCs, Week 12 (n = 42) | 3.97 (0.73)

10. Secondary Outcome: Mean Corpuscular Volume Levels Over Time
Description: Mean corpuscular volume (MCV) is a measure of the average red blood cell volume. MCV levels at Weeks -2, 4, 8, and 12 were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Mircera
Number analyzed (Participants) | 125
femtoliters
  MCV, Week -2 (n = 125) | 90.32 (7.32)
  MCV, Week 4 (n = 107) | 89.99 (7.53)
  MCV, Week 8 (n = 112) | 89.41 (7.04)
  MCV, Week 12 (n = 108) | 88.09 (8.79)

11. Secondary Outcome: Mean Values of Iron Parameters (Serum Iron and Total Iron Binding Capacity) Over Time
Description: Mean values of serum iron and total iron binding capacity (TIBC) were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microgram per deciliter
Arm/Group | Mircera
Number analyzed (Participants) | 131
microgram per deciliter
  Serum Iron, Week -2 (n = 131) | 102.13 (77.47)
  Serum Iron, Week 4 (n = 122) | 108.56 (59.65)
  Serum Iron, Week 8 (n = 118) | 116.79 (67.96)
  Serum Iron, Week 12 (n = 112) | 110.53 (56.31)
  TIBC, Week -2 (n = 131) | 273.44 (114.36)
  TIBC, Week 4 (n = 122) | 266.98 (116.69)
  TIBC, Week 8 (n = 115) | 283.50 (133.49)
  TIBC, Week 12 (n = 112) | 276.43 (118.54)

12. Secondary Outcome: Mean Values of Serum Ferritin Over Time
Description: Mean values of serum ferritin were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram per mililiter
Arm/Group | Mircera
Number analyzed (Participants) | 126
nanogram per mililiter
  Serum Ferritin, Week -2 (n = 126) | 1806.30 (6418.97)
  Serum Ferritin, Week 4 (n = 117) | 1422.48 (2550.43)
  Serum Ferritin, Week 8 (n = 109) | 1109.07 (1050.90)
  Serum Ferritin, Week 12 (n = 105) | 1109.80 (1016.17)

13. Secondary Outcome: Mean Values of Transferrin Over Time
Description: Mean values of transferrin were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: miligram per mililiter
Arm/Group | Mircera
Number analyzed (Participants) | 25
miligram per mililiter
  Transferrin, Week -2 (n = 25) | 168.24 (54.07)
  Transferrin, Week 4 (n = 16) | 160.00 (40.04)
  Transferrin, Week 8 (n = 18) | 165.72 (40.89)
  Transferrin, Week 12 (n = 18) | 159.22 (36.04)

14. Secondary Outcome: Mean Values of Transferrin Saturation Over Time
Description: Mean values of Transferrin Saturation (TSAT) were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Mircera
Number analyzed (Participants) | 125
Percentage
  TSAT, Week -2 (n = 125) | 45.55 (38.71)
  TSAT, Week 4 (n = 116) | 48.70 (36.31)
  TSAT, Week 8 (n = 109) | 46.08 (31.08)
  TSAT, Week 12 (n = 106) | 45.71 (29.81)

15. Secondary Outcome: Mean Values of Serum Albumin and Serum Globulin Over Time
Description: Mean values of serum albumin and serum globulin were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: gram per deciliter
Arm/Group | Mircera
Number analyzed (Participants) | 132
gram per deciliter
  Serum Albumin, Week -2 (n = 132) | 3.60 (0.53)
  Serum Albumin, Week 4 (n = 123) | 3.54 (0.42)
  Serum Albumin, Week 8 (n = 118) | 3.58 (0.46)
  Serum Albumin, Week 12 (n = 115) | 3.64 (0.46)
  Serum Globulin, Week -2 (n = 131) | 3.48 (0.65)
  Serum Globulin, Week 4 (n = 123) | 3.41 (0.68)
  Serum Globulin, Week 8 (n = 117) | 3.55 (0.73)
  Serum Globulin, Week 12 (n = 113) | 3.51 (0.67)

16. Secondary Outcome: Mean Values of Aspartate Aminotransferase, Alanine Transaminase and Serum Alkaline Phosphatase Over Time
Description: Mean values of aspartate aminotransferase (AST), alanine transaminase (ALT) and serum alkaline phosphatase were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units per litre
Arm/Group | Mircera
Number analyzed (Participants) | 131
units per litre
  AST, Week -2 (n = 128) | 23.48 (18.45)
  AST, Week 4 (n = 123) | 23.26 (12.87)
  AST, Week 8 (n = 117) | 22.86 (15.00)
  AST, Week 12 (n = 115) | 23.17 (15.69)
  ALT, Week -2 (n = 129) | 31.34 (27.52)
  ALT, Week 4 (n = 121) | 30.18 (18.82)
  ALT, Week 8 (n = 118) | 29.44 (20.26)
  ALT, Week 12 (n = 115) | 31.07 (20.71)
  Serum Alkaline Phosphatase, Week -2 (n = 131) | 154.7 (110.6)
  Serum Alkaline Phosphatase, Week 4 (n = 123) | 163.3 (108.9)
  Serum Alkaline Phosphatase, Week 8 (n = 118) | 162.1 (123.4)
  Serum Alkaline Phosphatase, Week 12 (n = 115) | 159.3 (100.1)

17. Secondary Outcome: Mean Values of Serum Creatinine, Blood Urea Nitrogen, Serum Phosphate and Serum Bilirubin Over Time
Description: Mean values of serum creatinine, blood urea nitrogen (BUN), serum phosphate and serum bilirubin were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: miligram per deciliter
Arm/Group | Mircera
Number analyzed (Participants) | 132
miligram per deciliter
  Serum Creatinine, Week -2 (n = 132) | 7.89 (2.96)
  Serum Creatinine, Week 4 (n = 123) | 8.34 (2.47)
  Serum Creatinine, Week 8 (n = 116) | 8.03 (2.36)
  Serum Creatinine, Week 12 (n = 115) | 8.19 (2.72)
  BUN, Week -2 (n = 131) | 57.72 (29.71)
  BUN, Week 4 (n = 122) | 60.67 (27.70)
  BUN, Week 8 (n = 117) | 60.10 (32.04)
  BUN, Week 12 (n = 113) | 61.79 (35.14)
  Serum Phosphate, Week -2 (n = 124) | 5.00 (4.70)
  Serum Phosphate, Week 4 (n = 114) | 5.02 (1.93)
  Serum Phosphate, Week 8 (n = 112) | 4.81 (1.64)
  Serum Phosphate, Week 12 (n = 107) | 5.37 (5.22)
  Serum Bilirubin, Week -2 (n = 131) | 0.52 (0.34)
  Serum Bilirubin, Week 4 (n = 123) | 0.50 (0.33)
  Serum Bilirubin, Week 8 (n = 118) | 0.52 (0.43)
  Serum Bilirubin, Week 12 (n = 115) | 0.51 (0.21)

18. Secondary Outcome: Mean Values of Serum Sodium and Serum Potassium Over Time
Description: Mean values of serum sodium and serum potassium were reported.
Time Frame: At Weeks -2, 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimole per liter
Arm/Group | Mircera
Number analyzed (Participants) | 132
millimole per liter
  Serum Potassium, Week -2 (n = 132) | 5.00 (0.94)
  Serum Potassium, Week 4 (n = 123) | 6.26 (11.74)
  Serum Potassium, Week 8 (n = 118) | 5.11 (0.88)
  Serum Potassium, Week 12 (n = 115) | 5.03 (1.08)
  Serum Sodium, Week -2 (n = 132) | 137.1 (4.36)
  Serum Sodium, Week 4 (n = 122) | 136.2 (12.65)
  Serum Sodium, Week 8 (n = 118) | 137.0 (4.58)
  Serum Sodium, Week 12 (n = 115) | 136.9 (5.37)

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: SAEs and non-serious AEs were reported for the safety population which included all participants who received at least one dose of study medication.
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 9/132
Other Adverse Events (participants affected / at risk) | 36/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=132)
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=132)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 4
Hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Peritoneal dialysis (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.